CLINICAL TRIAL: NCT03022929
Title: A Multifaceted Intervention to Improve Prescribing for Acute Respiratory Infection for Adults and Children in Emergency Department and Urgent Care Settings
Acronym: MITIGATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 986083; 971471 (Other: UC Davis IRB)
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapted Intervention (No Intervention): The investigators will use GetSmart materials published by the CDC appropriate to the emergency department and urgent care settings and select and adapt brochures and other campaign messages for acute care providers.
- Enhanced Intervention (Experimental): The investigators will use all of the methods of the Adapted Intervention. In addition to these methods, the investigators will add posters within exam rooms which will include modified GetSmart content and other nudges such as physician pictures with their signed public commitment to antibiotic stewardship or flair denoting commitment to stewardship. The investigators will also provide physicians with personalized monthly performance ranking with each physician receiving the designation of "top performer" or "not a top performer" based on their appropriate antibiotic prescribing practices for acute respiratory infections. This will be the Enhanced Antimicrobial Stewardship Commitment and Feedback intervention.
  Interventions: Behavioral: Enhanced Antimicrobial Stewardship Commitment and Feedback

INTERVENTIONS:
Behavioral: Enhanced Antimicrobial Stewardship Commitment and Feedback — Goes beyond the GetSmart recommendations to discern whether these recommendations can be improved upon.
  Arms: Enhanced Intervention

SUMMARY:
Inappropriate antibiotic use is a major public health concern. Excessive exposure to antibiotics results in emergence and spread of drug-resistant bacteria, potentially avoidable adverse drug reactions, and increased healthcare utilization and cost. As antibiotic prescribing in emergency departments and urgent care centers remains unchecked, national professional organizations including the Infectious Diseases Society of America (IDSA) and the Society for Healthcare Epidemiology (SHEA), and an Executive Order from the President of the United States, recommend expansion of antimicrobial stewardship to these ambulatory care settings. The goal of antimicrobial stewardship is to effectively promote judicious antibiotic use in all healthcare settings, yet stewardship programs have not achieved their potential in terms of either reach or effectiveness. Reach has been limited by implementation mostly in inpatient settings; at the same time, recent critical experiments in behavioral science suggest that the effectiveness of existing stewardship programs could be greatly augmented through inclusion of behavioral nudges, benchmarked audit and feedback, and peer-to-peer comparisons.

DETAILED DESCRIPTION:
In this proposed acute care project, the investigators will compare a package consisting of education for providers using existing materials from Center for Disease Control and Prevention's (CDC) GetSmart campaign adapted for the acute care setting led by a physician champion at each site (the adapted intervention), to a more intensive intervention that incorporates adapted GetSmart materials enhanced with individualized audit and feedback, peer comparisons, and behavioral nudges (the enhanced intervention). The comparative effectiveness of the enhanced intervention will be evaluated in a multicenter cluster randomized trial nested within a quasi-experimental study of acute care stewardship. The investigators' hypothesis is that both interventions will reduce inappropriate antibiotic prescribing for antibiotic nonresponsive acute respiratory infections (ARIs) in emergency departments and urgent care centers, but that the enhanced one will be more effective. The investigators will use an interrupted time series study design to measure the impact of their interventions against the baseline period of usual care as well as against seasonally-adjusted historical controls. The cluster randomized design for the two types of acute care stewardship interventions will allow measurement of the difference- in-differences in antibiotic prescribing rates for acute bronchitis, acute bronchiolitis, viral pharyngitis, influenza, and nonspecific upper respiratory infection (URI). Translation of proven behavioral techniques is a new and innovative approach to improving prescribing decisions. This project will expand stewardship to a new setting using innovative and effective approaches including the adaptation of behavioral techniques for emergency department (ED) and urgent care settings. The investigators will also further establish their research group as a network for developing novel tools, measuring outcomes for antimicrobial stewardship, and disseminating research findings through acute care setting-specific toolkits.

ELIGIBILITY:
Clinicians will be eligible for the study if they meet the following Inclusion Criteria:

1. Must be a clinician at one of the study sites.
2. Must treat adult and/or pediatric patients with an acute respiratory infections.

Individual patient encounters will be ineligible for analysis if they meet any of the following Exclusion Criteria:

1. Medical co-morbidities that make acute respiratory infection (ARI) guidelines less likely to apply.
2. Concomitant visit diagnoses indicating a non-ARI possible bacterial infection.
3. Concomitant visit diagnoses indicating potentially antibiotic appropriate ARI. diagnoses or other ARI diagnoses suggestive of a bacterial infection.
4. Visit occurred within 30 days of an earlier ARI diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2017-01; Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Antibiotic Prescribing Trends | Up to 2 years
  The investigators will measure the likelihood that an antibiotic is prescribed in an antibiotic-nonresponsive acute respiratory infection visit.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa S May, MD,MSPH,MSHS, Principal Investigator — Associate Professor and Director of Emergency Department Antibiotic Stewardship
Locations (3):
- United States (3):
  - UC Davis Medical Center, Sacramento, California
  - UCLA Harbor Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No
No IPD planned.